CLINICAL TRIAL: NCT02781675
Title: Effects of a Modified High-fat Mediterranean Dietary Pattern on Lipoprotein and Inflammatory Markers of CVD Risk in Adults
Brief Title: The Mediterranean Full-Fat Dairy Study
Acronym: MFFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-012
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Disease; Dyslipidemia; Inflammation
Keywords: Diet; Mediterranean; Cholesterol; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias; Inflammation | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Western Diet (Experimental): Dietary Intervention: 3 wks of a typical Western Diet
  Interventions: Other: Dietary Intervention
- Mediterranean Diet (Experimental): Dietary Intervention: 3 wks of a Mediterranean-style diet
  Interventions: Other: Dietary Intervention
- Modified Mediterranean Diet (Experimental): Dietary Intervention: 3 wks of a Mediterranean-style diet including full fat dairy products
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — 3 wk dietary intervention with prescribed menus and ~50% foods provided.

SUMMARY:
A Mediterranean dietary pattern emphasizing an abundance of plant-based foods including nuts, moderate intakes of fish, poultry and low-fat dairy products, and use of extra virgin olive oil as the main source of fat has been associated with reduced risk of cardiovascular disease (CVD), and such a pattern has been advocated by the 2015 U.S. Dietary Guidelines Advisory Committee. The strongest experimental support for this recommendation derives from the success of the recent PREDIMED CVD outcomes trial, and studies indicating that a Mediterranean-style diet improves lipoprotein and oxidative markers of cardiovascular disease risk in comparison to either low-fat or Western dietary patterns. However, in none of these studies were comparisons made between the effects of Mediterranean-style diets with low-/nonfat vs. full-fat dairy foods. The overall objective of the present proposal is to determine whether the inclusion of full-fat rather than low- and nonfat dairy foods in a Mediterranean dietary pattern based on that used in the PREDIMED study results in similar improvements in biomarkers of CVD risk. Specifically, we will test the hypotheses that 1) a standard Mediterranean diet will lower LDL-C and apoB compared to a Western diet; 2) modification of the Mediterranean diet by replacing low-fat dairy products with high-fat dairy (3 servings/day; high-dairy fat Mediterranean diet) will not significantly increase LDL-C and apoB but may raise large buoyant LDL particles compared with a standard Mediterranean diet; and 3) the high dairy fat and standard Mediterranean diets will result in comparable reductions in levels of inflammatory markers and oxidized LDL, and improvements in endothelial function compared to a Western diet.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35 kg/m2
* Weight stable for > 3 months
* Agrees to abstain from alcohol or dietary supplements during the study

Exclusion Criteria:

* History of coronary heart disease, cerebrovascular disease, peripheral vascular disease, bleeding disorder, liver or renal disease, diabetes, lung disease, HIV, or cancer (other than skin cancer) in the last 5 years.
* Current use of hormones or drugs knowns to affect lipid metabolism
* Use of nicotine products or recreational drugs
* Abnormal TSH
* Pregnant or breastfeeding
* Total- and LDL- cholesterol > 95th percentile for sex and age
* Fasting triglyceride > 500 mg/dl
* Fasting blood sugar > 126 mg/dl
* Blood pressure >160/95 mm Hg
* Allergy to or unwillingness to consume study foods

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Plasma LDL-cholesterol | 3 weeks
Plasma Apolipoprotein B | 3 weeks
Plasma Small LDL concentrations | 3 weeks
Plasma Large LDL particle concentrations | 3 weeks
Plasma Total LDL particle concentrations | 3 weeks

SECONDARY OUTCOMES:
Plasma triglycerides | 3 weeks
Plasma HDL-cholesterol | 3 weeks
Plasma apolipoprotein AI | 3 weeks
Plasma oxidized LDL | 3 weeks
Plasma C-reactive protein | 3 weeks
Plasma Interleukin-6 | 3 weeks
Plasma Intercellular Adhesion Molecule 1 (ICAM-1) | 3 weeks
Plasma Vascular Cell Adhesion Molecule 1 (VCAM-1) | 3 weeks
RH-PAT index (endothelial function) | 3 weeks
  Endothelial function measured by finger reactive hyperemia peripheral arterial tonography

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Cholesterol Research Center, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No